CLINICAL TRIAL: NCT05510141
Title: A Randomized Controlled Trial Comparing Virtual Reality Games Versus Nitrous Oxide for Pain Reduction in Common Outpatient Procedures in Pediatric Surgery
Brief Title: Virtual Reality Games in Pediatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Cordula Scherer, Dr.med, Insel Gruppe AG, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01446
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Analgesia; Surgical Procedure, Unspecified; Immersion
MeSH Terms: conditions — Agnosia | interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Gaming (Experimental)
  Interventions: Other: Virtual reality gaming
- Nitrous Oxide (Active Comparator): Standard procedure
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Other: Virtual reality gaming — Instead of nitrous oxide, which is the standard procedure, virtual reality gaming is applied to reach pain reduction in minor surgery procedures
  Arms: Virtual Reality Gaming
Drug: Nitrous oxide — Standard procedure
  Arms: Nitrous Oxide

SUMMARY:
Randomized controlled trial reporting the pain levels and pain control/reduction of children at the age of 6-15 undergoing surgical procedures by using virtual reality gaming (VR) compared to nitrous oxide. Therefore, 50 patients in each treatment group are recruited, resulting in 100 children altogether. The pain levels and pain control/reduction is measured by the standard anesthesia protocol normally used when nitrous oxide is applied and questionnaires that are administered to the patients at baseline and two weeks after surgery including both the primary and secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Indication to undergo an elective minor surgical procedure (removal of percutaneous osteosynthesis or pin material or dressing change)
* Written informed consent by parents
* Written informed consent by patient if patient is 14 or 15 years old

Exclusion Criteria:

* Inability to understand the VR-program
* Inability to fill in the questionnaire because of language deficiencies
* Neurologic disorders
* Respiratory tract infections
* Intolerance of the VR headset or VR gaming procedure

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual face scale of Bieri score directly after surgery | Directly after surgery (up to 20 minutes)
  Pain scale to measure pain reduction for children at the age 6-9, the score results in a pain score from 0-10 (0: minimum value, no pain; 10: maximum value, strongest imaginable pain)
Visual analogue scale (VAS) directly after surgery | Directly after surgery (up to 20 minutes)
  Pain scale to measure pain reduction for children at the age 11-15, the score results in a pain score from 0-10 (0: minimum value, no pain; 10: maximum value, strongest imaginable pain)
Visual face scale of Bieri score two weeks after surgery | Two weeks after surgery
  Pain scale to measure pain reduction for children at the age 6-9, the score results in a pain score from 0-10 (0: minimum value, no pain; 10: maximum value, strongest imaginable pain)
Visual analogue scale (VAS) two weeks after surgery | Two weeks after surgery
  Pain scale to measure pain reduction for children at the age 11-15, the score results in a pain score from 0-10 (0: minimum value, no pain; 10: maximum value, strongest imaginable pain)
Change in objective pain reaction measured by heart frequencies | During the procedure, estimated to be in average 15-20min
  Elevation of the heart rate indicates pain
Change in objective pain reaction measured by blood pressure | Before (up to 3 minutes) and directly after the surgery (up to 3 minutes)
  Elevation of blood pressure indicates pain, we measure the difference between the two measures

SECONDARY OUTCOMES:
Fun directly after surgery | Directly after surgery (up to 20 minutes)
  Did the patient have fun during the procedures, measured by questionnaires with a Likert Scale from 1 to 6 (1= no fun, 6= maximum of fun)
Fun two weeks after surgery | Two weeks after surgery
  Did the patient have fun during the procedures, measured by questionnaires with a Likert Scale from 1 to 6 (1= no fun, 6= maximum of fun)
Patient satisfaction directly after surgery | Directly after surgery (up to 20 minutes)
  The patient is asked in the questionnaires if he/she woud undergo the procedures again with a Likert Scale from 1 to 6 (1= would absolutely not do it again, 6= would absolutely do it again)
Patient satisfaction two weeks after surgery | Two weeks after surgery
  The patient is asked in the questionnaires if he/she woud undergo the procedures again with a Likert Scale from 1 to 6 (1= would absolutely not do it again, 6= would absolutely do it again)
Time limit of virtual reality gaming | During the surgery (estimated to be 3 to 25 minutes)
  The time is measured while nitrous oxide or virtual reality gaming is administered. The investigators evaluate if there is a time limit for virtual reality gaming, where they have to stop the intervention (comparable to the time limit of nitrous oxide application of 20 min)

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Scherer, Dr.med, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The final trial data set and statistical code will be made available from the corresponding author from three months following the final enrollment of patients within reasonable request, and will be published as mentioned in the ethical approvement. We plan to publish the study protocol in a peer-reviewed journal before end of enrolling.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Study Protocol: before end of enrolling Data Set and Statistical code: from three months following the final enrollment

REFERENCES:
- [Derived] Scherer C, Lanz LA, Liebs TR, Kaiser N, Zindel M, Berger SM. A randomized controlled trial comparing immersive virtual reality games versus nitrous oxide for pain reduction in common outpatient procedures in pediatric surgery. Trials. 2025 Jan 20;26(1):21. doi: 10.1186/s13063-025-08718-9. PMID 39833849